CLINICAL TRIAL: NCT01461590
Title: Phase II Trial of Transfusion Volumes in Children With Acute Severe Anaemia
Brief Title: Study of Safe Blood Transfusion Volumes to Correct Acute Severe Anaemia
Acronym: Tx30
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof Kathryn Maitland (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor-Investigator, Prof Kathryn Maitland, Professor in Infectious Diseases and Critical Care, KEMRI-Wellcome Trust Collaborative Research Program
Organization: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEMRI_CT_2011/0015
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Severe Anaemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20ml/kg of whole blood transfusion (Active Comparator): Standard care recommended by WHO
  Interventions: Other: Whole blood
- 30ml/kg of whole blood (Experimental): Higher volume than currently recommended
  Interventions: Other: Whole blood

INTERVENTIONS:
Other: Whole blood — 30mls/kg transfused over fours hours
Other: Whole blood — 20mls/kg transfused over four hours

SUMMARY:
Greater volume of whole blood(30mls/kg compared to 20mls/kg) following standard calculations, given to children with severe anaemia will be beneficial in haematological correction and can be given safely since respiratory distress and haemodynamic changes result from acidosis and compensation in these children rather than from biventricular failure.

DETAILED DESCRIPTION:
Severe anemia (SA, hemoglobin <6 g/dl) is a leading cause of pediatric hospital admission in Africa, with significant in-hospital mortality. The underlying etiology is often infectious, but specific pathogens are rarely identified. Guidelines developed to encourage rational blood use recommend a standard volume of whole blood (20 ml/kg) for transfusion, but this is commonly associated with a frequent need for repeat transfusion and poor outcome. Evidence is lacking on what haemoglobin threshold criteria for intervention and volume are associated with the optimal survival outcomes.

We evaluated the safety and efficacy of a higher volume of whole blood (30 ml/kg; Tx30: n = 78) against the standard volume (20 ml/kg; Tx20: n = 82) in Ugandan children (median age 35.5 months (interquartile range (IQR) 12.5 to 52.5)) for 24-hour anemia correction (hemoglobin >6 g/dl: primary outcome) and 28-day survival.

ELIGIBILITY:
Inclusion Criteria:

* Severe anaemia(HB less than 6g/dl)at admission
* Guardian or parent willing/able to provide consent

Exclusion Criteria:

* Malignancy
* Surgery
* Acute trauma
* Severe malnutrition

Ages: 60 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Correction of severe anaemia. | 24 hours
  Correction of severe anaemia to a Hb >6g/dL at 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Engoru, MMed, MBChB, Principal Investigator — Soroti Regional Hospital, Uganda
Locations (2):
- Uganda (2):
  - Mbale Regional Referral Hospital, Mbale, Mbale
  - Soroti Regional Hospital, Soroti, Soroti

REFERENCES:
- [Derived] Olupot-Olupot P, Engoru C, Thompson J, Nteziyaremye J, Chebet M, Ssenyondo T, Dambisya CM, Okuuny V, Wokulira R, Amorut D, Ongodia P, Mpoya A, Williams TN, Uyoga S, Macharia A, Gibb DM, Walker AS, Maitland K. Phase II trial of standard versus increased transfusion volume in Ugandan children with acute severe anemia. BMC Med. 2014 Apr 25;12:67. doi: 10.1186/1741-7015-12-67. PMID 24767094